CLINICAL TRIAL: NCT01226290
Title: Symptom Effectiveness Study of VizAblate™ Intrauterine Ultrasound-Guided RF Ablation (IUUSgRFA) in the Ablation of Uterine Fibroids
Brief Title: Fibroid Ablation Study
Acronym: FAST-EU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device changes; adequate enrollment achieved
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL02413
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Leiomyoma; Uterine Fibroids; Menorrhagia
Keywords: uterine fibroid RF ablation; intrauterine ultrasound; VizAblate
MeSH Terms: conditions — Leiomyoma; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VizAblate treatment (Experimental): VizAblate System: subject acts as her own control
  Interventions: Device: VizAblate System

INTERVENTIONS:
Device: VizAblate System — VizAblate enables a minimally invasive procedure to visualize, target, and ablate uterine fibroids using intrauterine ultrasound and radiofrequency (RF) energy.

SUMMARY:
The primary objective of this study is to establish the effectiveness and confirm the safety of the VizAblate System in ablating symptomatic uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* 28 years of age or older
* Regular, consistent menstrual cycles
* History of excessive bleeding
* One Menstrual Pictogram score ≥ 120 during a one-month screening period
* Baseline Uterine Fibroid Symptom & Quality of Life (UFS-QOL) Symptom Severity Subscale (SSS) score ≥ 20
* Between 1 and 5 Target Fibroids between 1 cm and 5 cm and/or maximum volume 82.4cc
* At least one fibroid must indent the endometrium
* Subject is not at material risk for pregnancy.
* Subject is willing to maintain use or non-use of hormonal contraception
* Subject is willing to have uniform maintenance (use or non-use) of any antifibrinolytic or nonsteroidal anti-inflammatory agents

Exclusion Criteria:

* Subserosal fibroids with bulk symptoms
* Presence of type 0 intracavitary fibroids
* Any Target Fibroid > 5 cm in maximum diameter with a volume > 82.4cc
* Any fibroid that obstructs access of the VizAblate probe
* Postmenopausal by history
* Desire for current or future fertility
* Hemoglobin < 6 g/dl
* Pregnancy
* Evidence of disorders of hemostasis
* Use of Gonadotropin-releasing hormone (GnRH) agonist or implantable or injectable progestin and/or estrogen, Selective Estrogen Receptor Modulators (SERM) or selective progesterone receptor modulator (SPRM)
* Short-term use of hormonal medication for management of bleeding
* Evidence for current cervical dysplasia
* Endometrial hyperplasia
* Confirmed abdominal / pelvic malignancy within the previous five years
* Active pelvic infection
* Clinically significant adenomyosis
* Previous uterine artery embolization. Previous surgical or ablative treatment for fibroids or menorrhagia within previous 12 months
* Current use of anticoagulant therapy
* Need for emergency surgery to treat fibroid symptoms
* Concomitant intrauterine polyps > 1.0 cm
* Contraindication to MRI
* Renal insufficiency
* Uncontrolled hypertension lasting 2 years or more
* One or more treatable fibroids that are calcified
* Chronic pelvic pain
* Presence of an extrauterine pelvic mass
* Presence of a tubal implant for sterilization
* Previous pelvic irradiation
* Endometrial cavity length < 4.5 cm

Min Age: 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in target fibroid perfused volume | 3 months

SECONDARY OUTCOMES:
Number of adverse events | procedure through 12 mo
  Procedure safety will be assessed by recording all adverse events that occur on the day of the procedure. Longer-term safety will be assessed by recording at each follow-up visit any untoward medical occurrence since baseline. Each adverse event will be assessed for severity and relationship to study device.
Percentage reduction in Menstrual Pictogram score | baseline through 12 months
Percentage reduction in the Symptom Severity Subscale (SSS) of the Uterine Fibroid Symptom and Quality of Life (UFS-QOL) questionnaire | baseline through 12 months
Rate of surgical reintervention for menorrhagia | through 12 months
Return to normal daily activity | 2 weeks or until returned to normal activity

OTHER OUTCOMES:
Subject satisfaction | 3 month, 6 month, 12 months
Anesthesia regimen | Day of procedure
System ease of use | End of study
Subject pain and tolerance of procedure | Day of procedure
HRQL sub scale of Uterine Fibroid Symptom Quality of Life (UFS-QOL) questionnaire | 3 month, 6 month, 12 months
EuroQOL EQ-5D | 3 month, 6 month, 12 month
Length of Stay | Day of procedure
Nonsurgical reintervention for menorrhagia | 30 day, 3 month, 6 month, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: David Toub, MD, Study Director — Gynesonics
Locations (10):
- Universidad Autonoma de Nuevo Leon (UANL), Monterrey, Nuevo León, Mexico
- Netherlands (4):
  - Máxima Medisch Centrum, Veldhoven, North Brabant
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Medisch Spectrum Twente, Enschede
- United Kingdom (5):
  - University College Hospital, London, London
  - Royal London Hospital, Whitechapel, London
  - Birmingham Women's NHS Foundation Trust, Birmingham, West Midlands
  - Princess Royal Hospital, Haywards Health, West Sussex
  - Bradford Teaching Hospitals NHS Trust, Bradford, West Yorkshire

REFERENCES:
- [Derived] Shifrin G, Engelhardt M, Gee P, Pschadka G. Transcervical fibroid ablation with the Sonata system for treatment of submucous and large uterine fibroids. Int J Gynaecol Obstet. 2021 Oct;155(1):79-85. doi: 10.1002/ijgo.13638. Epub 2021 Mar 17. PMID 33544889